CLINICAL TRIAL: NCT07089680
Title: Impact of Nirmatrelvir and Ritonavir (PAXLOVID®) on Mortality, Progression to Severe Disease, and Activities of Daily Living (ADL) Worsening in Long-term Care Hospitals (LTCHs) in Korea
Brief Title: A Study to Learn About the Study Medicine Paxlovid (Nirmatrelvir + Ritonavir) in Adults Aged 60 and Older Living in Korean Long-term Care Hospitals Who Have COVID-19
Status: Not yet recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4671064
Record Dates: First submitted 2025-07-24; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
Keywords: Nirmatrelvir / Ritonavir (Paxlovid); COVID-19; Activities of Daily Living (ADL); Long-Term Care Hospitals; Frailty
MeSH Terms: conditions — COVID-19; Frailty | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paxlovid treated group: Participants aged 60 years or older residing in long-term care hospitals (LTCHs) in Korea who were diagnosed with COVID-19 and received Paxlovid (Nirmatrelvir/Ritonavir) as part of their clinical care. This group will be assessed for multiple outcomes including mortality, progression to severe disease, worsening of activities of daily living (ADL), and frailty.
  Interventions: Drug: Nirmatrelvir/Ritonavir
- Paxlovid untreated group: Participants aged 60 years or older residing in long-term care hospitals (LTCHs) in Korea who were diagnosed with COVID-19 but did not receive Paxlovid treatment. This group serves as a comparator to evaluate the effectiveness of Paxlovid on outcomes such as mortality, progression to severe disease, ADL decline, and frailty.

INTERVENTIONS:
Drug: Nirmatrelvir/Ritonavir — Participants aged 60 years or older residing in long-term care hospitals (LTCHs) in Korea who were diagnosed with COVID-19 and received Paxlovid (Nirmatrelvir/Ritonavir) as part of their clinical care. This group will be assessed for multiple outcomes including mortality, progression to severe disease, worsening of activities of daily living (ADL), and frailty.
  Other Names: Paxlovid
  Groups: Paxlovid treated group

SUMMARY:
The purpose of this study is to learn about the effects of the study medicine (called Paxlovid) for the possible treatment of COVID-19 in older adults who live in long-term care hospitals (LTCHs) in Korea. Researchers want to know whether Paxlovid lowers the chance of severe illness or death and helps people carry out their usual daily activities, remain free from aging and weakness, and maintain cognitive function.

This study is seeking participants who:

* are 60 years of age or older
* live in a long-term care hospital in Korea
* were diagnosed with COVID-19 on or after 14 January 2022, during the period when Paxlovid was available as part of routine care
* received Paxlovid within 5 days after their first COVID-19 symptoms (only for people in the Paxlovid group)

All participants in this study received their usual COVID-19 care. About half also received Paxlovid. Paxlovid was prescribed as part of routine care at the long-term care hospital, typically taken by mouth 2 times a day for 5 days.

The study team will compare the health results of people who received Paxlovid to those who did not, using similar parameters such as age, sex, and medical history. This will help the study team to understand whether Paxlovid makes a meaningful difference in stopping severe illness, death, or slow-down daily functioning.

Participants will not have any extra study visits or tests. The study team will only review information already recorded in their medical charts for up to 1 year after their COVID-19 symptom onset.

ELIGIBILITY:
1. LTCH residents ≥60 years of age, diagnosed with COVID-19 via SARS-CoV-2 PCR or antigen test, with a symptom onset date (index date) between 14 January 2022 and 1 June 2023 (or latest date available)
2. Dispensed Paxlovid within 5 days of COVID-19 symptom onset (Paxlovid treated patients only)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes residents of long-term care hospitals (LTCHs) in Korea who are aged 60 years or older and were diagnosed with COVID-19 between January 14, 2022 and June 1, 2023 (or latest available date). Diagnosis was confirmed by SARS-CoV-2 PCR or antigen test, and symptom onset date was available. Participants were either treated with Paxlovid (Nirmatrelvir/Ritonavir) within 5 days of symptom onset or received no antiviral treatment. Patients were excluded if they received other COVID-19 treatments (e.g., remdesivir, molnupiravir, monoclonal antibodies), had severe renal or hepatic dysfunction, or had contraindicated medications. The study uses retrospective medical chart data and includes follow-up for up to 365 days.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of progression to severe disease or all-cause mortality within 30 days | During index date, defined as 30 days from COVID-19 symptom onset. Index period: 14 Jan 2022 to 1 June 2025 (or latest date available)

SECONDARY OUTCOMES:
Change in Activities of Daily Living (ADL) from baseline at 30 days | During index date, defined as 30 days from COVID-19 symptom onset. Index period: 14 Jan 2022 to 1 June 2025 (or latest date available)
Change in Activities of Daily Living (ADL) from baseline at 90 days | During index date, defined as 30 days from COVID-19 symptom onset. Index period: 14 Jan 2022 to 1 June 2025 (or latest date available)
Change in Activities of Daily Living (ADL) from baseline at 365 days | During index date, defined as 30 days from COVID-19 symptom onset. Index period: 14 Jan 2022 to 1 June 2025 (or latest date available)
All Cause mortality at 30 days by baseline ADL dependency | During index date, defined as 30 days from COVID-19 symptom onset. Index period: 14 Jan 2022 to 1 June 2025 (or latest date available)
Progression to severe disease at 30 days by baseline ADL dependency | During index date, defined as 30 days from COVID-19 symptom onset. Index period: 14 Jan 2022 to 1 June 2025 (or latest date available)
ADL change at 30 days by baseline ADL dependency | During index date, defined as 30 days from COVID-19 symptom onset. Index period: 14 Jan 2022 to 1 June 2025 (or latest date available)
Subgroup analysis of ADL change at 90 days by baseline ADL dependency | During index date, defined as 30 days from COVID-19 symptom onset. Index period: 14 Jan 2022 to 1 June 2025 (or latest date available)
Subgroup analysis of ADL change at 365 days by baseline ADL dependency | During index date, defined as 30 days from COVID-19 symptom onset. Index period: 14 Jan 2022 to 1 June 2025 (or latest date available)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.